CLINICAL TRIAL: NCT00039676
Title: Clinical, Laboratory, and Epidemiologic Characterization of Individuals and Families at High Risk of Blood and Lymph Node Malignancy
Brief Title: Clinical, Laboratory and Epidemiologic Characterization of Individuals and Families at High Risk of Hematologic Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020210; 02-C-0210; NCT00052234 (obsolete NCT alias)
Record Dates: First submitted 2002-06-06; First posted 2002-06-07 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-28

CONDITIONS: Waldenstrom Macroglobulinemia; Chronic Lymphocytic Leukemia; Hodgkin Disease; NonHodgkin Lymphoma; Mixed Lymphoproliferative Disease
Keywords: Genetics; Risk Factors; Natural History; Lymphoma; Leukemia; Lymph Node Cancer
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma; Leukemia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard: People that have blood or lymph node cancer, or a family history of leukemia or lymphoma.

SUMMARY:
Background:

* Individuals may be prone to develop blood or lymph node cancers (leukemia or lymphoma) for a variety of reasons, including genetic predisposition to these cancers, environmental exposures or other medical conditions.
* Studies of people and families at high risk of cancer often lead to clues about their cause that may also be important regarding the sporadic occurrence of these cancers in the general population.
* Identifying genetic or environmental factors that play a role in the development of these diseases may be important in developing prevention trials, screening programs and treatments.

Objectives:

* Describe the cancers and other conditions in families with blood or lymph node cancer.
* Find and describe genes that may cause blood and lymph node cancer, and understand how they work in families.
* Use laboratory methods to try to determine if it is possible to identify who is at highest risk of blood or lymph node cancer.
* Test how genes act with other factors to alter the risk of disease, its severity or its manifestations in families.

Eligibility:

* Individuals of any age with a personal or family history of a blood or lymph node cancer.
* Individuals with a personal or family history of medical conditions or environmental exposures that may predispose to blood or lymph node cancer.

Design:

* Participants complete questionnaires about their personal and family medical history and provide consent for researchers to review their medical records and pathology materials related to their care and those of deceased relatives with blood or lymph node cancer, tumors, or other related illnesses for whom they are the legally authorized representative.
* Participants donate a sample of blood or cheek cells, or a lock of hair for genetic studies.
* Patients may also be evaluated at the NIH Clinical Center by one or more of the following specialists: cancer doctor or blood specialist, medical geneticist, research nurses or clinical social worker. They may have blood and urine tests and a cheek swab or mouth wash to collect cheek cells. Some patients may also be asked to have x-rays and routine imaging, such as CT scans or ultrasound tests, cell surface markers, skin biopsy, and, with special consents, bone marrow biopsy, MRI or PET scans, apheresis or fluorescein angiography and photography.

DETAILED DESCRIPTION:
Background:

Persons may be prone to develop hematologic or lymphoproliferative cancer for a variety of reasons including: inherited predisposition of benign, premalignant, or malignant conditions; environmental exposures shared by family members; previous tumors or preneoplastic conditions; immune deficiency; or stochastic processes

Investigations of individuals and families at high risk of cancer often lead to etiologic clues that may be important in the sporadic counterparts of these cancers in the general population

Identification of etiologically important genetic factors could inform chemoprevention trials, screening programs, and treatment of hematologic and lymphoproliferative cancers

Objectives:

To evaluate and define the clinical spectrum and natural history of disease in syndromes predisposing to hematologic cancer

To evaluate potential precursor states of malignancy in families at risk

To quantify the risks of specific tumors in family members and define syndromic constellations

To identify, map, characterize, clone, and determine function of tumor susceptibility genes

To validate and test associations of biomarkers with risk

To identify genetic determinants, environmental factors, and gene-environmental interactions conferring cancer risk in individuals and families

To identify differences and similarities between the familial and sporadic condition

To educate and counsel study participants about their risk of hematologic malignancy including prevention recommendations and early detection activities when known

To develop syndrome-specific educational materials for medical professionals and high-risk family members

Eligibility:

On referral, persons >= 11 months will be included only because of personal history, and persons >/=18 years can also be included because of personal or family history of the parameters listed below:

* a medical history of hematologic/lymphoproliferative malignancy of an unusual type, pattern, or number or
* there are known or suspected factor(s) predisposing to hematologic malignancy, either genetic or congenital factors, environmental exposure, or unusual demographic features

  * For familial neoplasms, two or more living affected cases among family members are generally required

Design:

This is a prospective study. Families are studied long-term using a cohort approach.

The study design and evaluation vary by the specific type of familial neoplasm being studied

The overall approach to eligible families includes defining affection status, characterization of disease, localization of genetic loci, identification of genes, evaluation of phenotype/genotype correlations, estimation of risk of the disease associated with carrier

status and identification of other risk factors that modify penetrance (genetic, environmental, and host factors)

ELIGIBILITY:
* INCLUSION CRITERIA:

On referral, persons >= 11 months will be included only because of personal history, and persons >=18 years can also be included because of personal or family history of the parameters listed below:

* A medical history of hematologic/ lymphoproliferative malignancy of an unusual type, pattern, or number or
* Known or suspected factor(s) predisposing to hematologic malignancy, either genetic and/or congenital factors (birth defects, metabolic phenotype, chromosomal anomalies or Mendelian traits associated with tumors), environmental exposure (medications, occupation, radiation, diet, infectious agents, etc.), or unusual demographic features (very young age of onset, multiple tumors, etc.)

Personal and family medical history must be verified through questionnaires, interviews, and review of pathology slides and medical records. For familial neoplasms, two or more living affected cases among family members are generally required, although in selected instances exceptions may be made, e.g., for WM, one case plus a living 1st degree relative with an autoimmune condition will qualify a family for further investigations.

Disease-specific considerations. Familial aggregation of any hematologic cancer(s) is eligible for study. Disease-specific procedures are outlined in appendices:

1. Chronic lymphocytic leukemia (CLL)
2. Waldenstrom macroglobulinemia (WM)
3. Non-Hodgkin lymphoma (NHL)
4. Hodgkin lymphoma (HL)
5. Mixed/miscellaneous hematologic and lymphoproliferative diseases

Ability of subject or Legally Authorized Representative (LAR) to understand, and the willingness to sign, a written informed consent document.

EXCLUSION CRITERIA:

* Referred individuals for whom reported diagnoses cannot be verified;
* Referred individuals who decline informed consent.

Min Age: 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: General population with a family history of cancer
Sampling Method: Non-Probability Sample
Enrollment: 1836 (Actual)
Dates: Start 2002-07-08 (Actual)

PRIMARY OUTCOMES:
Clinical Spectrum and Natural History | Ongoing
  To define the clinical spectrum and natural history of familial blood and lymph node malignancies and susceptibility states over time.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Stewart, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - NIH National Cancer Institute - Shady Grove, Rockville, Maryland

REFERENCES:
- [Background] Berndt SI, Camp NJ, Skibola CF, Vijai J, Wang Z, Gu J, Nieters A, Kelly RS, Smedby KE, Monnereau A, Cozen W, Cox A, Wang SS, Lan Q, Teras LR, Machado M, Yeager M, Brooks-Wilson AR, Hartge P, Purdue MP, Birmann BM, Vajdic CM, Cocco P, Zhang Y, Giles GG, Zeleniuch-Jacquotte A, Lawrence C, Montalvan R, Burdett L, Hutchinson A, Ye Y, Call TG, Shanafelt TD, Novak AJ, Kay NE, Liebow M, Cunningham JM, Allmer C, Hjalgrim H, Adami HO, Melbye M, Glimelius B, Chang ET, Glenn M, Curtin K, Cannon-Albright LA, Diver WR, Link BK, Weiner GJ, Conde L, Bracci PM, Riby J, Arnett DK, Zhi D, Leach JM, Holly EA, Jackson RD, Tinker LF, Benavente Y, Sala N, Casabonne D, Becker N, Boffetta P, Brennan P, Foretova L, Maynadie M, McKay J, Staines A, Chaffee KG, Achenbach SJ, Vachon CM, Goldin LR, Strom SS, Leis JF, Weinberg JB, Caporaso NE, Norman AD, De Roos AJ, Morton LM, Severson RK, Riboli E, Vineis P, Kaaks R, Masala G, Weiderpass E, Chirlaque MD, Vermeulen RCH, Travis RC, Southey MC, Milne RL, Albanes D, Virtamo J, Weinstein S, Clavel J, Zheng T, Holford TR, Villano DJ, Maria A, Spinelli JJ, Gascoyne RD, Connors JM, Bertrand KA, Giovannucci E, Kraft P, Kricker A, Turner J, Ennas MG, Ferri GM, Miligi L, Liang L, Ma B, Huang J, Crouch S, Park JH, Chatterjee N, North KE, Snowden JA, Wright J, Fraumeni JF, Offit K, Wu X, de Sanjose S, Cerhan JR, Chanock SJ, Rothman N, Slager SL. Meta-analysis of genome-wide association studies discovers multiple loci for chronic lymphocytic leukemia. Nat Commun. 2016 Mar 9;7:10933. doi: 10.1038/ncomms10933. PMID 26956414
- [Background] Rotunno M, McMaster ML, Boland J, Bass S, Zhang X, Burdett L, Hicks B, Ravichandran S, Luke BT, Yeager M, Fontaine L, Hyland PL, Goldstein AM; NCI DCEG Cancer Sequencing Working Group; NCI DCEG Cancer Genomics Research Laboratory; Chanock SJ, Caporaso NE, Tucker MA, Goldin LR. Whole exome sequencing in families at high risk for Hodgkin lymphoma: identification of a predisposing mutation in the KDR gene. Haematologica. 2016 Jul;101(7):853-60. doi: 10.3324/haematol.2015.135475. Epub 2016 Jun 13. PMID 27365461
- [Background] Goldin LR, McMaster ML, Rotunno M, Herman SE, Jones K, Zhu B, Boland J, Burdett L, Hicks B, Ravichandran S, Luke BT, Yeager M, Fontaine L, Goldstein AM, Chanock SJ, Tucker MA, Wiestner A, Marti G, Caporaso NE. Whole exome sequencing in families with CLL detects a variant in Integrin beta 2 associated with disease susceptibility. Blood. 2016 Nov 3;128(18):2261-2263. doi: 10.1182/blood-2016-02-697771. Epub 2016 Sep 14. No abstract available. PMID 27629550
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-C-0210.html